CLINICAL TRIAL: NCT03000374
Title: Preoperative Induction Therapy With 12 Weeks of Panitumumab in Combination With mFOLFOX-6 in an Enriched Population (Quadruple Wild-Type) of Patients With mrT3 Rectal Cancer of the Middle Third With Clear Mesorectal Fascia
Brief Title: Induction Therapy With Panitumumab + mFOLFOX-6 in Rectal Cancer and Quadruple Wild-type Mutation Before Surgery
Acronym: PIER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Collaborators: Pivotal S.L. (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD-1601; 2016-002333-29 (EudraCT Number)
Record Dates: First submitted 2016-11-14; First posted 2016-12-22 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Panitumumab; Fluorouracil; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Panitumumab + mFOLFOX-6 (Experimental): - Modified FOLFOX-6 regimen: 5-Fluorouracil (5-FU), oxaliplatin and leucovorin will be administered intravenously once every 14 days, according to the mFOLFOX-6 regimen:
  Day 1: Oxaliplatin 85 mg/m² in IV infusion of 250-500 mL and leucovorin 200 mg/m² IV, both injected over two hours, followed by 5-FU 400 mg/m2 in IV bolus and a 46-hour infusion of 5-FU 2400 mg/m².
  - Panitumumab will be administered intravenously (IV) in a dose of 6 mg/kg on day 1 every 14 days. Panitumumab will be supplied to sites by the study sponsor in 5-mL and 20-mL vials, at a concentration of 20 mg/mL.
  Treatment will continue until 6 cycles have been administered, followed by surgery, 5 weeks +/- 1 week after the last dose of neoadjuvant treatment
  Interventions: Drug: Panitumumab; Drug: 5Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin

INTERVENTIONS:
Drug: Panitumumab — Panitumumab will be administered intravenously (IV) in a dose of 6 mg/kg on day 1 every 14 days. Panitumumab will be supplied to sites by the study sponsor in 5-mL and 20-mL vials, at a concentration of 20 mg/mL.
  Other Names: Vectibix 20 mg/ml
Drug: 5Fluorouracil — Once every 14 days. Day 1: 400 mg/m2 in IV bolus and a 46-hour infusion of 5-FU 2400 mg/m².
  Other Names: 5-FU
Drug: Oxaliplatin — Once every 14 days. Day 1: 85 mg/m2 I.V. infusión in 250-500 mL, over two hours, followed by 5-FU
  Other Names: Any marketed
Drug: Leucovorin — Once every 14 days. Day 1: 200 mg/m2 I.V., over two hours, followed by 5-FU
  Other Names: Any marketed

SUMMARY:
Patients with rectal adenocarcinoma of intermediate risk (defined by magnetic resonance imaging [MRI]), without mutations in KRAS, BRAF, NRAS and PI3KCA, who are candidates for preoperative treatment, will receive a preoperative Induction therapy with 12 weeks of panitumumab with mFOLFOX-6 to evaluate the efficacy in terms of pathologic complete response (pCR)

DETAILED DESCRIPTION:
Phase II, nonrandomized single-arm trial of preoperative treatment with mFOLFOX-6 and panitumumab in an enriched population of patients with rectal adenocarcinoma of intermediate risk, screened by MRI, without mutations in KRAS, BRAF, NRAS and PI3K. All patients enrolled in the study will receive 12 weeks of the investigational product (mFOLFOX-6 with panitumumab) every 14 days for six cycles, unless unacceptable toxicity occurs or progression is detected. After this treatment, response will be evaluated by diffusion-weighted MRI and endoscopy. In the absence of disease progression, patients eligible for R0 resection will undergo total mesorectal excision (TME). After surgery, patients will receive mFOLFOX6 x 6 cycles. In the case of intolerance to FOLFOX-panitumumab, disease progression or ineligibility for R0 resection, patients will receive chemoradiotherapy with capecitabine 825 mg/m2 every 12 hours concomitantly with radiotherapy (RT) with a total dose of 50.4 Gy. At the end of this treatment, patients will undergo TME between 6-8 weeks after finishing the CRT. If a patient has received 4 or more neoadjuvant cycles of FOLFOX-panitumumab before unacceptable toxicity or progression, it will be considered that the neoadjuvant treatment has been completed and the patient will have no additional neoadjuvant treatment but surgery. If the patient has received <4 cycles of neoadjuvant treatment, neoadjuvant CRT will be administered.

If a patient has an acceptable toxicity or disease progression or a R0 surgery is not possible to be performed and the patient received CRT, the patient will be followed up for 24 months, from the enrollment of the last patient in the trial, or until progression occurs, in order to assess progression-free survival and all the data regarding surgery and CRT will be recorded in the eCRF. If a patient withdraws consent and refuses to continue participating in the study, follow-up evaluations must be discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form, and willingness and ability to comply with the requirements of the protocol;
2. Men or women with rectal cancer, age ≥ 18 and <75 years;
3. Histologically documented adenocarcinoma of the rectum. All other histologic types are excluded. A biopsy of the rectal primary tumor must be available (between 1-4), with tumor representation > 50% in each sample. The samples will be sent to Val d'Hebron Institute of Oncology (VHIO) for molecular determination. The blocks of the biopsies will be sent included in paraffin.
4. Rectal cancer candidate for R0 resection with preservation of the rectal sphincter.
5. Tumors with the following characteristics on high-resolution thin-slice (3 mm) MRI:

   1. mrT3
   2. Tumors of the middle third, defined as tumors whose distal edge is ≤ 12 cm of the anal verge or below the peritoneal reflection and above ≥ 2 cm of the anorectal junction.
   3. Absence of MRF invasion, defined as a distance ≥ 1 mm between the tumor and the fascia;
6. Absence of mutations in KRAS (mutations in KRAS exon 2 [codons 12/13], exon 3 [codons 59/61] and exon 4 [codon 117/146], NRAS (NRAS exon 2 [codons 12/13], exon 3 [codons 59/61] and exon 4 [codons 117/146]), BRAF (exon 15 [codon 600] and PI3KCA in exons 9 and 20
7. ECOG performance status ≤ 2;
8. Hematological status:

   * Neutrophils (ANC) ≥ 1.5 x 109/L;
   * Platelets ≥ 100 x 109/L;
   * Hemoglobin ≥ 9 g/dL;
9. Adequate renal function: serum creatinine <1.5 x upper limit of normal (ULN);
10. Adequate liver function:

    * Serum bilirubin ≤ 1.5 x ULN,
    * Alkaline phosphatase < 5 x ULN,
    * AST/ALT < 3 x ULN;
11. Regular monitoring feasible;
12. In women of childbearing potential, a negative serum pregnancy test within 1 week (7 days) before the start of study treatment;
13. Women must commit to using reliable and appropriate methods of contraception for up to at least six months after the end of the study treatment (when applicable). Men with a partner of childbearing potential must agree to use a method of contraception and their partners must use another contraceptive method for the duration of the trial. Sexual abstinence will be accepted as a contraception method, with the duration and considerations stablished by the investigator

Exclusion Criteria:

1. Mucinous adenocarcinoma.
2. N2 lymph node involvement, defined as: 4 or more lymph nodes in the mesorectum showing morphological signs of metastatic involvement on MRI. A lymph node is considered malignant when:

   1. Short axis > 9 mm.
   2. Short axis 5-9 mm and ≥2 of the following criteria:

      i Rounded appearance. ii Heterogeneous margin. iii Heterogeneous signal intensity.
   3. Short axis < 5 mm AND round shape AND heterogeneous margin AND heterogeneous signal intensity.
3. Extramesorectal lymph node involvement: an involved extramesorectal lymph node is defined as a lymph node in the obturator area with a short axis > 8 mm, round shape and heterogeneous signal..
4. Prior treatment with panitumumab or cetuximab;
5. Preexisting permanent neuropathy (grade ≥ 2 NCI-CTCAE);
6. Concomitant antitumor treatment not foreseen in the protocol (e.g., chemotherapy, targeted molecular therapy, immunotherapy);
7. Treatment with any other investigational medicinal product within the 28 days prior to study entry;
8. Other simultaneous or prior malignancy, except: i) properly treated uterine cervix carcinoma in situ, ii) basal or squamous cell skin carcinoma, iii) cancer in complete remission for a period > 5 years;
9. Evidence of metastatic disease in additional studies or in the physical examination;
10. Any other severe and uncontrolled nonmalignant disease, major surgery or traumatic injury in the last 28 days;
11. Pregnant or breastfeeding women;
12. Patients with known allergy to any excipient of the investigational products;
13. Clinically significant cardiovascular disease, including myocardial infarction, unstable angina, symptomatic congestive heart failure or cardiac arrhythmia in the year before randomization in the study.
14. Intestinal occlusion: In the case of intestinal occlusion, patients may be enrolled in the study after performing a derivative stoma.
15. Interstitial Lung Disease

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | Up to 16-18 weeks after first treatment administration
  Pathologic CR is defined as the absence of viable tumor cells in the primary tumor and lymph nodes (ypT0N0).

SECONDARY OUTCOMES:
Rates of R0 resection and free mesorectal fascia (or circumferential margin) | Up to 16-18 weeks after first treatment administration
Tumor regression grade (TRG) | Up to 16-18 weeks after first treatment administration
  the residual tumor after preoperative treatment is evaluated semi-quantitatively using the 5-point regression grading scale established by Dworak
Rate of tumor downstaging (mrT versus ypT) | Up to 16-18 weeks after first treatment administration
Quality of surgery | Up to 16-18 weeks after first treatment administration
  According to the histopathology report
Adverse events and changes in laboratory results | All AEs that occur up until 30 days after the last dose of investigational product will be recorded. Serious and nonserious AEs related with the study treatment that appear up until 30 days after the administration of the last dose should be reported.
  The adverse events will be encoded using the Medical Dictionary for Regulatory Activities (MedDRA), version 18.1 or later, and evaluated using the U.S. National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 4.0.
Surgical complications | Over 30 days after surgery.
Rate of local recurrence | At 3 years after recruitment
Distant metastasis rate | At 3 years after recruitment
Disease free survival | At 3 years after recruitment
Overall survival | At 3 years after recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Fernández-Martos, MD, Study Director — Initia Centro Oncológico Integral
Locations (11):
- Spain (11):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital de Sabadell, Sabadell, Barcelona
  - Hospital de Sant Joan Despí Moisés Broggi, Sant Joan Despí, Barcelona
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No